CLINICAL TRIAL: NCT01844934
Title: Impact of Prehabilitation in Total Knee Arthroplasty: Outcomes and Healthcare Service Utilization
Brief Title: Impact of Prehabilitation in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Laura Franco, Physical therapist, Allina Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Study 3963-2 IRB
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Knee Arthroplasty; Knee Replacement; Prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: 2 arms, one intervention, one control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (No Intervention): The no intervention group will receive standard treatment that includes a four hour class pre-surgery consisting of a description of the surgery, what to expect in the hospital and during recovery and some exercises to be done in preparation for surgery.
- Prehabilitation (Experimental): Prehabilitation:The experimental group will receive a three week prehabilitation program prior to surgery in addition to standard treatment.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — The three week, 3 days / week prehabilitation exercise program will consist of resistance training, step training and stretching(flexibility) as well as cardiovascular endurance training. Intensity of training will increase over the three weeks. Classes will be delivered over a four week period with a gap during the third week allowing additional time for participants to practice their exercises. The home exercise program will be designed to account for the additional week.
  Arms: Prehabilitation

SUMMARY:
A study comparing the benefits of pre-habilitation exercise to standard care prior to total knee arthroplasy

DETAILED DESCRIPTION:
Recovery post Total Knee Replacement Surgery ((TKA) has been a subject of interest. In a study of 379 patients who had hip or knee replacement surgery, it was reported that at 6 months post-surgery patients with better baseline function had superior functional ability and less pain than patients with lower function at baseline. Another study of 276 patients undergoing TKA reported that pre-operative joint function was a predictor of joint function and overall function at 6 months post-surgery. These findings suggest that prehabilitation to increase functional ability prior to TKA may have a positive effect in recovering post-surgery. In a randomized control trial of patients receiving TKA, the group receiving an Exercise Program (prehabilitation) made significant improvements in performance from baseline to before surgery, and at 1 and 3 months post surgery. For the group that did not receive the Exercise Program pre-surgery, significant improvement did not occur until 3 months post surgery. The overall objective of the proposed single-blinded randomized controlled trial is to demonstrate that a well designed prehabilitation program for patients receiving TKA surgery will significantly improve outcomes related to pain and function and may reduce utilization of health care services post surgery.

In this randomized control trial we hypothesize that the group of participants who receive a prehabilitation Exercise Program will recover quicker than patients who do not receive the Exercise Program based on several measures of performance including pain, quadriceps strength, range of motion and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo unilateral TKA surgery
* Ambulatory
* Community dwelling (living at home)
* Able to participate in moderate intensity exercise
* American Society of Anesthesiologists Physical Status Classification(ASA) 1 - 3
* Speaks English

Exclusion Criteria:

* Patients who are planning a second surgery of the lower limbs during the six months post-surgery
* Have the effect of peripheral vascular disease or stroke on walking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from baseline to pre-surgery, 4, 14 and 26 weeks post surgery
  WOMAC, a self-assessment tool, is a valid and reliable instrument developed specifically to measure outcomes related to interventions for treatment of the hip and knee. Consisting of three domains: physical, pain and stiffness; a total score is derived by aggregating the domain scores.

SECONDARY OUTCOMES:
Six Minute Walk | Change from baseline to pre-surgery, 4, 14, 26 weeks post-surgery
  A valid and reliable measure of total distance walked in six minutes.
Gait Speed | Change from baseline to pre-surgery, 4, 14 and 26 weeks post surgery
  Gait speed will be measured with the 10 meter walk. It will be assessed under two conditions: 1) instructed to walk at normal speed, 2) instructed to walk as fast as possible.
Knee Range of Motion (ROM) | Change from baseline to pre-surgery, 4, 14, and 26 weeks post surgery
  Knee ROM (extension and flexion) will be measured with a goniometer at the surgical joint.
Medical Outcomes Study Short Form-36 (SF-36) | Change from baseline to pre-surgery, 4, 14 and 26 weeks post surgery
  The SF-36 measures 8 dimensions of outcome: physical functioning, social functioning, role-physical, bodily pain, mental health, role-emotional, vitality and general health.
Sit-to-stand repetitions in 30 seconds | Change from baseline to pre-surgery, 4, 14 and 26 weeks post surgery
  Number of complete stand up to sit down cycles is counted.
Pain | Change from baseline to pre-surgery, 4, 14 and 26 weeks post surgery
  Pain will be measured upon completion of each of the functional tasks (gait speed, six-minute walk and sit to stand) using a Visual Analog Scale from 0 to 10 where 0 is no pain and 10 is severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Crandall, M.D., Principal Investigator — Unity Hospital, Allina Health; Laura Franco, PT, OCS, Principal Investigator — Courage Kenny Rehabilitation Institute, Allina Health
Locations (1):
- Unity Hospital, Fridley, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No